CLINICAL TRIAL: NCT00808249
Title: A Multi-Center, Randomized, Placebo-Controlled, Double-Blind, Parallel Group, Efficacy and Safety Study of AZD7325 in the Treatment of Generalized Anxiety Disorder (GAD)
Brief Title: AZD7325 Proof of Concept in Patients With Generalized Anxiety Disorder (GAD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark A. Smith, MD PhD, Medical Science Director, Emerging Psychiatry, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1140C00006
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Results first posted 2011-05-19 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2011-04

CONDITIONS: Anxiety Disorders
Keywords: Generalized Anxiety Disorder; GAD; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder | interventions — 4-amino-8-(2-fluoro-6-methoxy-phenyl)-N-propylcinnoline-3-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (4):
- A-AZD7325 2mg (Experimental): AZD7325 2mg BID
  Interventions: Drug: AZD7325
- B-AZD7325 5mg (Experimental): AZD7325 5mg BID
  Interventions: Drug: AZD7325
- C-AZD7325 10mg (Experimental): AZD7325 10mg QD
  Interventions: Drug: AZD7325
- D-Placebo (Experimental): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD7325 — 2 tablets taken twice a day for 28 days
  Arms: A-AZD7325 2mg
Drug: AZD7325 — 2 tablets taken twice a day for 28 days
  Arms: B-AZD7325 5mg
Drug: AZD7325 — 2 tablets taken twice a day for 28 days
  Arms: C-AZD7325 10mg
Drug: Placebo — 2 tablets taken twice a day for 28 days
  Arms: D-Placebo

SUMMARY:
The purpose of this research study is to determine whether AstraZeneca's drug AZD7325 is safe and effective in the treatment of generalized anxiety disorder.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent before any study-related procedures start.
* The patient is previously diagnosed with Generalized Anxiety Disorder.
* The patient has a HADS-A (anxiety) score ≥10 at both screening and randomization.

Exclusion Criteria:

* Patient has a lifetime history of schizophrenia or other psychotic disorders
* Patient has a history of seizures or seizure disorder.
* Patient is pregnant or breast feeding.
* Patient has received electroconvulsive treatment (ECT) in the past.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 725 (Actual)
Dates: Start 2008-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A. Smith, MD, PhD, Study Director — AstraZeneca; David V. Sheehan, Principal Investigator — University of South Florida College of Medicine
Locations (52):
- United States (52):
  - Research Site, Birmingham, Alabama
  - Research Site, Tucson, Arizona
  - Research Site, Arcadia, California
  - Research Site, Beverly Hills, California
  - Research Site, Cerritos, California
  - Research Site, Chino, California
  - Research Site, Encino, California
  - Research Site, Los Alamitos, California
  - Research Site, Novato, California
  - Research Site, Oceanside, California
  - Research Site, San Diego, California
  - Research Site, Norwich, Connecticut
  - Research Site, Fort Myers, Florida
  - Research Site, Miami, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Saint Petersberg, Florida
  - Research Site, Tampa, Florida
  - Research Site, Winter Park, Florida
  - Research Site, Atlanta, Georgia
  - Research Site, Marietta, Georgia
  - Research Site, Smyrna, Georgia
  - Research Site, Libertyville, Illinois
  - Research Site, Park Ridge, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Overland Park, Kansas
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Cambridge, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Clementon, New Jersey
  - Research Site, Fresh Meadows, New York
  - Research Site, Mount Kisco, New York
  - Research Site, New York, New York
  - Research Site, Rochester, New York
  - Research Site, Raleigh, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Bismarck, North Dakota
  - Research Site, Beechwood, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Middleburg Heights, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Portland, Oregon
  - Research Site, Jenkintown, Pennsylvania
  - Research Site, Norristown, Pennsylvania
  - Research Site, Memphis, Tennessee
  - Research Site, Friendswood, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Salt Lake City, Utah
  - Research Site, Woodstock, Vermont
  - Research Site, Herndon, Virginia
  - Research Site, Spokane, Washington
  - Research Site, Middleton, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: International multi-center study, 44 sites recruited between Dec 2008 and May 2009
Pre-assignment Details: Screening for eligibility and wash-out of restriced medications. 725 subjects enrolled but 424 subjects were randomized. Number of participants analyzed is the number of subjects in MITT (modified intent to treat) population, it is different with any of population listed in the participant flow chart.
Groups:
- A-AZD7325 2 mg: AZD7325 2 mg BID
- B-AZD7325 5 mg: AZD7325 5 mg BID
- C-AZD7325 10 mg: AZD7325 10 mg QD
Period: Overall Study
Arm/Group | A-AZD7325 2 mg | B-AZD7325 5 mg | C-AZD7325 10 mg | D-Placebo
Started | 107 | 106 | 105 | 106
Completed | 90 | 91 | 83 | 90
Not Completed | 17 | 15 | 22 | 16
Not completed — Adverse Event | 4 | 7 | 10 | 6
Not completed — Lost to Follow-up | 2 | 3 | 3 | 5
Not completed — Withdrawal by Subject | 4 | 0 | 2 | 4
Not completed — Protocol Violation | 3 | 3 | 3 | 0
Not completed — Lack of Efficacy | 1 | 1 | 0 | 0
Not completed — study specific discontinuation criteria | 1 | 0 | 1 | 0
Not completed — All other reasons | 2 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A-AZD7325 2 mg | B-AZD7325 5 mg | C-AZD7325 10 mg | D-Placebo | Total
Number analyzed (Participants) | 107 | 106 | 105 | 106 | 424
Age, Customized [Number; unit: Participants]
  18-39 | 44 | 43 | 48 | 53 | 188
  40-65 | 63 | 63 | 57 | 53 | 236
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 62 | 61 | 62 | 247
  Male | 45 | 44 | 44 | 44 | 177

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Hamilton Rating Scale for Anxiety (HAM-A) Total Score
Description: The HAM -A is a 14-item clinician administered scale for the evaluation of anxiety symptoms. Each HAM-A item is rated on a 0 (not present) to 4 (very severe) scale, higher score indicates high level of anxiety. The HAM-A total score is calculated as the sum of 14 individual scores, with 56 as the maximum.
Time Frame: From randomization (baseline) to week 4
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | A-AZD7325 2 mg | B-AZD7325 5 mg | C-AZD7325 10 mg | D-Placebo
Number analyzed (Participants) | 105 | 105 | 103 | 102
Units on scale | -10.9 (0.87) [lower limit 0.87] | -11.1 (0.86) [lower limit 0.86] | -11.5 (0.87) [lower limit 0.87] | -10.9 (0.88) [lower limit 0.88]

2. Secondary Outcome: Change in Hospital Anxiety and Depression Scale for Anxiety (HADS-A) Total Score
Description: The HADS-A is a 7 item, self administered instrument to measure level of anxiety. Each item is a score rate from 0 (happens rarely ) to 3 (happens frequently), and the items are totaled for a maximum score of 21. The mimimum score 0 indicates that the patient rarely suffered from anxiety symptoms.
Time Frame: From randomization (baseline) to week 4
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | A-AZD7325 2 mg | B-AZD7325 5 mg | C-AZD7325 10 mg | D-Placebo
Number analyzed (Participants) | 105 | 105 | 103 | 102
Units on scale | -4.5 (0.49) [lower limit 0.49] | -4.2 (0.49) [lower limit 0.49] | -5.2 (0.50) [lower limit 0.50] | -4.6 (0.50) [lower limit 0.50]

3. Secondary Outcome: Change in Psychic Anxiety Symptoms as Measured by HAM-A Psychic Anxiety Factor Score
Description: The HAM-A psychic anxiety factor score is calculated as the sum of 7 HAM-A individual items related with psychic anxiety ( each rated from 0 to 4, 0 is the best). The minimum score for HAM-A psychic anxiety factor is 0 and maximum score is 28, higher score indicates severe psychic anxiety symptoms.
Time Frame: From baseline (randomization) to week 4
Measure: Least Squares Mean (Standard Error); unit: Unit on scale
Arm/Group | A-AZD7325 2 mg | B-AZD7325 5 mg | C-AZD7325 10 mg | D-Placebo
Number analyzed (Participants) | 105 | 105 | 103 | 102
Unit on scale | -5.9 (0.51) [lower limit 0.51] | -5.8 (0.51) [lower limit 0.51] | -6.5 (0.52) [lower limit 0.52] | -5.8 (0.52) [lower limit 0.52]

4. Secondary Outcome: Change in Somatic Symptoms as Measured by HAM-A Somatic Factor Score
Description: The HAM-A somatic factor score is calculated as the sum of 7 individual HAM-A items (each is rated from 0 to 4, 0 is the best) related with somatic anxiety symptoms. The minimum score for HAM-A somatic factor is 0 and maximum score is 28, higher score indicates severe somatic anxiety symptoms
Time Frame: From baseline ( randomization) to week 4
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | A-AZD7325 2 mg | B-AZD7325 5 mg | C-AZD7325 10 mg | D-Placebo
Number analyzed (Participants) | 105 | 105 | 103 | 102
Units on scale | -5.0 (0.41) [lower limit 0.41] | -5.3 (0.41) [lower limit 0.41] | -5.1 (0.42) [lower limit 0.42] | -5.2 (0.42) [lower limit 0.42]

5. Secondary Outcome: Change in Sheehan Disability Scale (SDS) Global Total Score
Description: The Sheehan Disability Scale is a patient-rated measure of functional disability in 3 subscales: work, social, and family life. Each subscale is rated from 0 to 10, with 0 as the best. SDS global total score is calculated as the sum of 3 subscales and ranges from 0(unimpaired) to 30 (highly impaired)
Time Frame: From baseline ( randomization) to week 4
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | A-AZD7325 2 mg | B-AZD7325 5 mg | C-AZD7325 10 mg | D-Placebo
Number analyzed (Participants) | 81 | 78 | 75 | 81
Units on scale | -4.7 (0.79) [lower limit 0.79] | -5.7 (0.80) [lower limit 0.8] | -6.8 (0.82) [lower limit 0.82] | -6.8 (0.79) [lower limit 0.79]

ADVERSE EVENTS:
Description: Number at risk is number of patients in safety population. The participant flow shows patients randomized and completed the study. The numbers are not the same since 2 patients were randomized but did not take study drug.
Arm/Group | A-AZD7325 2 mg | B-AZD7325 5 mg | C-AZD7325 10 mg | D-Placebo
Serious Adverse Events (participants affected / at risk) | 1 | 1 | 0 | 0
Other Adverse Events (participants affected / at risk) | 13 | 18 | 32 | 14
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | A-AZD7325 2 mg | B-AZD7325 5 mg | C-AZD7325 10 mg | D-Placebo
Road Traffic Accident (Injury, poisoning and procedural complications) | 0/106 | 1/106 | 0/105 | 0/105
Grand Mal Convulsion (Nervous system disorders) | 0/106 | 1/106 | 0/105 | 0/105
Anxiety (Psychiatric disorders) | 1/106 | 0/106 | 0/105 | 0/105
Deep Vein Thrombosis (Vascular disorders) | 1/106 | 0/106 | 0/105 | 0/105
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | A-AZD7325 2 mg | B-AZD7325 5 mg | C-AZD7325 10 mg | D-Placebo
Dizziness (Nervous system disorders) | 13/106 | 18/106 | 32/105 | 12/105
Headache (Nervous system disorders) | 8/106 | 17/106 | 9/105 | 14/105
Sedation (Nervous system disorders) | 5/106 | 6/106 | 10/105 | 1/105
Somnolence (Nervous system disorders) | 13/106 | 9/106 | 17/105 | 6/105
Euphoric Mood (Psychiatric disorders) | 7/106 | 11/106 | 10/105 | 6/105
Insomnia (Psychiatric disorders) | 4/106 | 5/106 | 2/105 | 7/105
Dry Mouth (Gastrointestinal disorders) | 6/106 | 4/106 | 11/105 | 7/105
Fatigue (General disorders) | 8/106 | 7/106 | 5/105 | 3/105
Feeling Abnormal (General disorders) | 1/106 | 4/106 | 8/105 | 0/105
Nausea (Gastrointestinal disorders) | 10/106 | 9/106 | 10/105 | 8/105

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other